CLINICAL TRIAL: NCT07182955
Title: Determinants of Cardiorespiratory Fitness and Effects of High Intensity Interval Training (HIIT) in Patients With Angina and No Obstructive Coronary Artery Disease (ANOCA)
Brief Title: Determinants of Cardiorespiratory Fitness and Effects of HIIT in Patients With ANOCA Obstructive Coronary Artery Disease(ANOCA)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Jamieson Bourque, MD, Professor of Medicine & Radiology, Medical Director of Nuclear Cardiology and Stress Laboratory, Medical Director of Echocardiography, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 302240
Record Dates: First submitted 2025-07-11; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: MINOCA; Shortness of Breath; Atherosclerotic Heart Disease of Native Coronary Artery
Keywords: ANOCA/MINOCA; High Intensity Interval Training; CPET Phenotype; Cardiorespiratory Fitness
MeSH Terms: conditions — MINOCA; Dyspnea | interventions — Exercise; Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): Remote 4 weeks of high-intensity interval exercise training on three non-consecutive days of the week.
  Interventions: Behavioral: EXERCISE TRAINING WITH OR WITHOUT MEDICATION

INTERVENTIONS:
Behavioral: EXERCISE TRAINING WITH OR WITHOUT MEDICATION — Remote 4 weeks of high-intensity interval exercise training on three non-consecutive days of the week.

SUMMARY:
The main goal is to understand what causes reduced fitness in ANOCA and whether targeted exercise can help improve it.

This study aims to better understand why patients with Angina and No Obstructive Coronary Artery Disease (ANOCA) have poor cardiorespiratory fitness and its effect on quality of life.

Investigators also want to see if a structured high-intensity exercise program (HIIT), done with remote monitoring, can safely improve heart function, fitness, and quality of life in these patients. The Investigators will use a special exercise test called cardiopulmonary exercise testing to look for patterns that can help explain exercise limitations and quality of life in ANOCA before and after a remote high-intensity exercise program.

DETAILED DESCRIPTION:
The overall research plan is for 25 subjects with angina and no obstructive coronary artery disease (ANOCA) on invasive or coronary CT angiography (ANOCA Study Population) to undergo cardiopulmonary exercise testing (CPET) to assess exercise workload and hemodynamic variables and health-related quality of life (HRQOL) measurement at baseline, followed by repeat testing after high-intensity interval exercise training for 4 weeks. The investigators will examine the diagnostic role of exercise by determining the relationship between exercise fitness and assessing the degree of cardiac, ventilatory, and muscle impairment on CPET.

Anginal burden and related functional status will be assessed via the Seattle Anginal Questionnaire. Overall functional status will be assessed through the Short form (SF36) and MacNew forms, levels of cardiac anxiety through the Cardiac Anxiety Questionnaire (CAQ), and effects on work absenteeism and presenteeism through the Work Limitations Questionnaire (WLQ). Baseline exercise status will be documented through the Duke Activity Status Index form.

The investigators will identify cardiorespiratory fitness peak oxygen consumption (VO2peak) and CPET phenotype with ANOCA. The investigators hypothesize that patients with ANOCA will have reduced VO2 peak and heterogeneous CPET phenotypes with substantial and varying contributions of cardiac, ventilatory, and muscle impairment. Phenotyping of determinants of exercise intolerance will be carried out using the following CPET parameters: cardiac-VO2peak, non-invasive cardiac output with CO2 rebreathing, and O2pulse; ventilatory via VE/VO2and oxygen uptake efficiency slope (OUES); muscle by VE/VCO2 slope, a-vO2 difference, and quadriceps muscle strength on isokinetic dynamometry. The Investigators predict that cardiac impairment will be the most frequent CPET phenotype in ANOCA, and this group will have poor exercise fitness.

The investigators will perform a 4-week high-intensity interval exercise training in 25 patients with ANOCA. The investigators will examine the feasibility of a remote exercise program with ramp exercise thresholds. The investigators predict that exercise program session adherence will be >80% based on preliminary data. The investigators will assess the effect of HIIT on CPET phenotype, improvement in VO2peak in patients with varying CPET phenotypes, model entropy, and HRQOL overall score and specific functional domains. The investigators predict that VO2peak will significantly improve with HIIT.

The exercise protocol for subjects will entail one initial supervised exercise session. All subsequent exercises will be done remotely. Each heart rate monitor will be programmed with heart rate zones that are 85-90% of that subject's angina threshold on the CPET. Subjects will be instructed to start with one 1-minute exercise and one 1-minute rest. The protocol will increase the length of exercise with the goal of getting up to four 4-minute sessions of exercise on three non-consecutive days of the week.

Remote HIIT will be accomplished using Polar heart rate monitoring and the Polar flow application. Patients will receive one supervised, treadmill exercise training session with all other exercise sessions performed remotely (brisk walking).

Participants will be provided with a wrist-based Polar Unite, which measures movement as well as heart rate (green LED) and transmits data to a centralized Polar storage site. Participants will be asked to wear the Polar device every day during the study. In addition, during intervention sessions, participants will be asked to wear the chest stripe to get a more accurate recording of HR to follow the exercise prescription.

Study staff will help set up the Polar watch and Polar Application and will demonstrate how to use them. Subjects will be given one training session in the exercise physiology core lab in which they will be shown how to follow the exercise regimen via their Polar device and also shown how to properly use the equipment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85
* ANOCA (Anginal symptoms of chest pain or exertional dyspnea suspected to be from myocardial ischemia Invasive or CT coronary angiogram without obstructive epicardial CAD (≥50% left main or ≥70% other epicardial stenosis or fractional flow reserve ≤0.80)
* Able to use the wearable and participate in a remote exercise program
* Able to participate in intermittent high-intensity training.
* Able to perform cardiopulmonary exercise testing (CPET)
* Able to provide Health-related quality of life questionnaire (HRQOL)
* Participants must be able to understand and provide informed consent in English and complete the study questionnaire in English

Exclusion Criteria:

* Systolic heart failure (LVEF <50% or NYHA class III symptoms)
* Prior myocardial infarction, coronary revascularization
* Inability to safely undergo cardiopulmonary exercise testing, based on investigator's judgment
* Pregnancy (due to unknown effects on CPET exercise markers)
* Inability to provide informed consent
* Life expectancy <1 year
* Prisoners
* Cognitively impaired
* Non-English speaking

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-04-14 (Estimated)

PRIMARY OUTCOMES:
Examine cardiorespiratory fitness (change in VO2max in mL/kg/min) with cardiopulmonary exercise testing (CPET) Phenotype. | 4 weeks
  The investigators will assess VO2max (mL/kg/min) in 25 patients with ANOCA at the exercise laboratory.

SECONDARY OUTCOMES:
Assess Changes in cardio-respiratory fitness (CRF) (VO2max) with High-Intensity Interval Exercise Training (HIIT) in Patients with ANOCA. | 4 weeks
  The investigators will examine the feasibility of a remote exercise program using ramp exercise thresholds. Based on preliminary data, they predict that adherence to the exercise sessions will exceed 80%. After four weeks of remote exercise, the investigators will reassess cardiorespiratory fitness (VO2max in mL/kg/min) after the HIIT intervention.
Health Related Quality Of Life (HRQOL) questionnaire | 4 Weeks
  The investigators will assess the health-related quality of life at baseline, alongside exercise testing, and again four weeks after the completion of the study to evaluate any changes.

CONTACTS AND LOCATIONS:
Overall Officials: Jamieson M Bourque, MD, MHS, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Angadi SS, Jarrett CL, Sherif M, Gaesser GA, Mookadam F. The effect of exercise training on biventricular myocardial strain in heart failure with preserved ejection fraction. ESC Heart Fail. 2017 Aug;4(3):356-359. doi: 10.1002/ehf2.12149. Epub 2017 Mar 16. PMID 28772048
- [Background] Hambrecht R, Walther C, Mobius-Winkler S, Gielen S, Linke A, Conradi K, Erbs S, Kluge R, Kendziorra K, Sabri O, Sick P, Schuler G. Percutaneous coronary angioplasty compared with exercise training in patients with stable coronary artery disease: a randomized trial. Circulation. 2004 Mar 23;109(11):1371-8. doi: 10.1161/01.CIR.0000121360.31954.1F. Epub 2004 Mar 8. PMID 15007010